CLINICAL TRIAL: NCT03190473
Title: The OPTIMIZE Trial to Assess the Procedural and Clinical Value of the Svelte IDS and RX Sirolimus Eluting Coronary Stent Systems for the Treatment of Atherosclerotic Lesions in a Randomized Study
Brief Title: OPTIMIZE IDE for the Treatment of ACS
Acronym: OPTIMIZE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company financial insolvency, not due to safety or efficacy concerns
Sponsor: Svelte Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IP-15-001
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Svelte (Experimental)
  Interventions: Device: DES
- Control (Active Comparator)
  Interventions: Device: DES

INTERVENTIONS:
Device: DES — PCI with implantation of a DES

SUMMARY:
Indication for use: "The Svelte DES is indicated for improving coronary luminal diameter in patients with symptomatic heart disease, including patients with non-ST elevation MI due to discrete de novo native coronary artery lesions. The treated lesion length should be less than the nominal stent length with a reference vessel diameter of 2.25 mm - 4.00 mm

ELIGIBILITY:
Inclusion Criteria:

* Subject is an eligible candidate for percutaneous coronary intervention (PCI);
* Subject has symptomatic coronary artery disease with objective evidence of ischemia or silent ischemia;
* Subject is an acceptable candidate for coronary artery bypass grafting (CABG);
* Subject has up to 3 de novo target lesions in up to 2 native coronary artery vessels, with no more than 2 lesions in a single vessel, each meeting the angiographic criteria and none of the exclusion criteria.
* Target lesion(s) must be located in a native coronary artery with a visually estimated reference vessel diameter (RVD) ≥ 2.25 mm and ≤ 4.00 mm;

Exclusion Criteria:

* The subject has cardiogenic shock, hemodynamic instability requiring inotropic or mechanical circulatory support, intractable ventricular arrhythmias, or ongoing intractable angina;
* The subject's target lesion(s) is located in the left main artery;
* The subject's target lesion(s) is located within 3 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCX) coronary artery by visual estimate;
* The subject's target lesion(s) is located within a saphenous vein graft or arterial graft;
* The subject's target lesion(s) will be accessed via a saphenous vein graft or arterial graft;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1630 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months

SECONDARY OUTCOMES:
Target Vessel Failure (TVF) | 6 and 12 months, and annually through 5 years
Major Adverse Cardiac Event (MACE) | 6 and 12 months and annually through 5 years follow-up
Stent Thrombosis | 6 and 12 months and annually through 5 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Shing C Wong, MD, Study Director — Svelte Medical
Locations (72):
- United States (54):
  - Thomas Hospital, Fairhope, Alabama
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Bakersfield Memorial Hospital, Bakersfield, California
  - Mission Cardiovascular Research Institute (Washington Hospital), Fremont, California
  - Long Beach VA Medical Center, Long Beach, California
  - Keck Hospital of USC, Los Angeles, California
  - San Francisco VA, San Francisco, California
  - Christiana Hospital, Newark, Delaware
  - Morton Plant Hospital, Clearwater, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - University of Miami Medical Center, Miami, Florida
  - Mediquest (Munroe Regional Medical Center), Ocala, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Jesse Brown VAMC, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Amita/Adventist Heart and Vascular, Hinsdale, Illinois
  - Elkhart General Healthcare, Elkhart, Indiana
  - St Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Mercy Hospital Medical Center, Des Moines, Iowa
  - Union Memorial Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Borgess Heart Center, Kalamazoo, Michigan
  - Northern Michigan Hospital d.b.a McLaren Northern Michigan, Petoskey, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Mary's Duluth Clinic, Duluth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - North Mississippi Health Services, Tupelo, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - NYU Winthrop Hospital, Mineola, New York
  - NYU Langone Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - St. Joseph's Hospital Health Center, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Durham VA Medical Center, Durham, North Carolina
  - Moses Cone Memorial Hospital, Greensboro, North Carolina
  - North Carolina Heart and Vascular, Raleigh, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Hershey Medical Center, Hershey, Pennsylvania
  - Robert Packer Hospital, Sayre, Pennsylvania
  - Texas Heart Institute, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Austin Heart, Round Rock, Texas
  - South Texas Cardiology Institute, San Antonio, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Swedish Hospital Medical Center, Seattle, Washington
- Japan (9):
  - Shonan Kamakura General Hospital, Kamakura
  - Kanazawa Cardiovascular Hospital, Kanazawa
  - Kokura Memorial Hospital, Kitakyushu
  - Medical Corporation Association Sakura Association Takahashi Hospital, Kobe
  - Ohara Healthcare Foundation Kurashiki Central Hospital, Kurashiki
  - Shin Koga Hospital, Kurume
  - Miyazaki Medical Association, Miyazaki
  - The Sakakibara Heart Institute of Okayama, Okayama
  - Sapporo Higashi Tokushukai Hospital, Sapporo
- Netherlands (9):
  - Meander Medisch Centrum, Amersfoort
  - OLVG loc Oost, Amsterdam
  - Tergooi Ziekenhuis, Blaricum
  - Amphia Ziekenhuis, Breda
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Catharina Ziekenhuis, Eindhoven
  - St Antonius Ziekenhuis, Nieuwegein
  - HAGA Ziekenhuis, The Hague
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kereiakes DJ, Feldman RL, Ijsselmuiden AJJ, Saito S, Amoroso G, Zidar JP, Wong SC, Stella P, Yakubov S, Lasala J, Cohen DJ, Doros G, Cutlip DE, Rao SV. Safety and Effectiveness of the SVELTE Fixed-Wire and Rapid Exchange Bioresorbable-Polymer Sirolimus-Eluting Coronary Stent Systems for the Treatment of Atherosclerotic Lesions: Results of the OPTIMIZE Randomized Study. Circ Cardiovasc Interv. 2021 Sep;14(9):e010609. doi: 10.1161/CIRCINTERVENTIONS.121.010609. Epub 2021 Aug 6. PMID 34353122
- [Derived] Mauri L, Doros G, Rao SV, Cohen DJ, Yakubov S, Lasala J, Wong SC, Zidar J, Kereiakes DJ. The OPTIMIZE randomized trial to assess safety and efficacy of the Svelte IDS and RX Sirolimus-eluting coronary stent Systems for the Treatment of atherosclerotic lesions: Trial design and rationale. Am Heart J. 2019 Oct;216:82-90. doi: 10.1016/j.ahj.2019.07.003. Epub 2019 Jul 13. PMID 31415994